CLINICAL TRIAL: NCT03000153
Title: Goals in Mind: A Randomised Controlled Evaluation of the Effectiveness of Tracking Goals in Counselling
Brief Title: Effectiveness of Tracking Goals in Counselling
Acronym: Goals in MIND
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Organisational changes at site meant that recruitment was no longer feasible.
Sponsor: University of Roehampton (Other)
Collaborators: MIND Tower Hamlets (Unknown)
Responsible Party: Principal Investigator, Mick Cooper, Professor of Counselling Psychology, University of Roehampton
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSYC 16/ 251
Record Dates: First submitted 2016-12-17; First posted 2016-12-21 (Estimated); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: Mental Health Impairment

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Completing the Goals Form (Experimental): In this arm, client participants will complete the Goals Form in collaboration with their therapists at the start of every session.
  Interventions: Other: Completing the Goals Form
- therapy as usual (No Intervention): In this arm, clients will have therapy as usual.

INTERVENTIONS:
Other: Completing the Goals Form — The Goals Form is a personalised outcome measure where clients enter their goals in collaboration with their assessor. Goals are then rated at the start of every session and open the therapeutic dialogue.
  Other Names: Goals Form
  Arms: Completing the Goals Form

SUMMARY:
Recent evidence suggests that focusing on positive goals rather than problems to avoid, may be associated with better psychological health and attainment of goals. In addition, the advantages of using personalised measures have been highlighted in a number of studies. The Goals Form is a new measure that comprises both elements. It invites clients, in collaboration with their therapist, to identify up to seven goals for therapy typically at a first assessment session and then to rate them on a 1-7 Likert scale, with 1 being not at all achieved and 7 being completely achieved. This research is important for clinical practice as it provides the foundations to identify what might be a helpful factor in counselling and psychotherapy.

The aim of the study is to test whether the use of the Goals Form leads to better clinical outcomes in counselling and psychotherapy. Participants in this study are counsellors and service users at Tower Hamlets Mind. The design of this study is a trial, which looks at comparing outcome measure scores in 'therapy as usual' and 'therapy using the Goals Form' when participants are randomly assigned to one of the two conditions. Interventions in this study involve using the Goals Form at the start of every session and taking part in a 30 minute interview once therapy has ended to give feedback about using the form in therapy . In addition to assessing outcome, the study also serves to compare satisfaction scores across the two conditions. It is a pilot to determine the feasibility of such trial including recruitment rates over a period of a year, adherence of counsellors and clients to the protocol, and the ethical issues raised.

DETAILED DESCRIPTION:
In recent years, there has been a rapid rise in the use of outcome and feedback measures in the counselling and psychotherapy field. In part, this is because evidence suggests that the systematic collection and integration of client feedback improves outcome across client populations, professional discipline, and model used. In a meta-analysis of five trials comparing use of a routine feedback protocol with treatment as usual (TAU) for adults receiving individual psychotherapy, there were significant gains for feedback groups over TAU, especially for clients identified as at risk for premature dropout or negative outcomes (Lambert, 2010). In a review of studies using the Partners for Change Outcome Monitoring system, clients using brief outcome measures at each session were 3.5 times more likely to experience reliable change and had half the odds of deterioration than those in TAU (Duncan, 2010, 2011; Lambert & Shimokawa, 2011; Murphy & Duncan, 2010). Currently, three randomized, controlled trials indicate improved outcomes using this system (Anker, Duncan, & Sparks, 2009; Reese, Norsworthy, & Rowlands, 2009; Reese, Toland, Slone, & Norsworthy, 2010). Based on the overall strength of current evidence, Lambert and Shimokawa (2011, p. 72) recommended that 'clinicians seriously consider making formal methods of collecting client feedback a routine part of their daily practice'.

At present, most psychological measurement is conducted using nomothetic scales. These are based on questions chosen by professional experts and consisting of checklists of symptoms (e.g., CORE-OM, PHQ-9). These questions are selected to be acceptable to large populations. However, given the diversity of problems presenting to mental health care services, a more personalised approach to psychological measurement might seem appropriate. Such an approach would shift the emphasis of measurement away from predefined, professionally-driven criteria, replacing it with a focus on those criteria given importance by the individual client. Individualised measures are questionnaires that include questions which can be generated by clients alone or in collaboration with the practitioner. This results in clients creating their own tailor-made questionnaire which only contains items that have meaning for them. Items are rated for intensity in a similar procedure to that of standardised measures.

The advantages of using individualised measures have been highlighted in a number of studies (e.g., Ashworth et al., 2005). Client-generated measures are evidenced to be user-friendly as individuals themselves identify areas of personal concern. Clinical improvement therefore, is evaluated according to topics of relevance to the individuals concerned. Research indicates that the fact that people themselves identify their own personal problems or goals which are meaningful to them and which reflect their individual needs, leads to more engagement in therapy (Turner-Stokes, 2011). Also, individualised measures are flexible and take into account the client's idiosyncratic variables such as personality, socioeconomic status and cultural background (Sales & Alves, 2012).

However, to date, the most commonly used personalised measures, such as the Personal Questionnaire (Elliott et al., 2015) and the PSYCHLOPS (Ashworth et al., 2005), focus on clients' difficulties rather than their goals. Research suggests that this may be problematic: there is evidence to suggest that focusing on positive goals to approach, rather than negative problems to avoid, may be associated with better psychological health and attainment of goals (Elliot & Church, 2002; Elliot & Friedman, 2007).

Hence, the aim of this study is to evaluate the benefits, to both the process and outcomes of therapy, of using a personalised goal form: the Goals Form. The Goals Form (Appendix 2.1) is an individualised outcome measure used to assess attainment of personal objectives for therapy. It was used as part of an initial open-label trial of pluralistic therapy (Cooper et al., 2015), and invites clients, in collaboration with their therapist, to identify up to seven goals for therapy typically at a first assessment session and then to rate them on a 1 7 Likert scale, with 1 being not at all achieved and 7 being completely achieved (Cooper, 2014). The agreed goals are then typed onto a digital copy of the form and printed off, such that the client is able to rate the same goals at regular intervals, ideally every session. Over the course of therapy, clients may choose to delete, add or modify goals, and the electronic copy of the Goals Form is revised accordingly. The Goals Form has shown satisfactory levels of internal reliability, and convergent validity against CORE-10, GAD-7 and PHQ-9. It is also sensitive to change in clinical populations (Cooper, 2014; Michael, Cooper, & Fugard, 2015).

In terms of user acceptability, clients' gave the Goals Form a mean rating of 4.2 on a 5-point helpfulness scale (SD = 1.2, n = 17), with a median and modal rating of 5 (very helpful). Ten of the 17 respondents (58.8%) gave it this highest rating. By contrast, the mean rating of the PHQ-9 was 3.7 (SD = 1.0, n = 17), with a median and modal rating of 4 (helpful). Intro to change interview (Cooper et al., 2015). In terms of why the Goals Form was helpful, five interviewees in Cooper et al.'s (2015) study said that it gave them a sense of progress, both from session to session and over the course of therapy. Interviewee 1, for instance, said: 'It kind of gave me a barometer on what I was doing'. Five of the participants said that it gave focus and structure to the therapy, reminding them of what they had come to work on and 'where you want to be at the end' (Interviewee 10). Interviewee 6, for instance, said: 'I'm a very scatty mind…because I was very depressed I couldn't concentrate and then it's helpful to have something in black and white on paper because then you knew this is what you were working at.' Two of the interviewees said the Goals Form was helpful because it encouraged them to reflect on how they had gone about achieving their objectives, and one said that they had felt challenged by it. In terms of negative aspects of the Goals Form, two participants said that they did not feel that they were good at naming goals, particular at the start of their therapy. Two of the interviewees said that they had been confused by the constant changes in goals, and one said that they felt the form needed to be explained more clearly.

Aims:

The objective of this study is to evaluate the impact of identifying and monitoring goals in therapy on clinical outcomes.

Hypothesis:

Client allocated to a goals-oriented condition will show significantly greater clinical improvement than clients in a standard counselling condition.

Procedure:

Clients will be allocated to counsellors as per standard clinic protocols. Clients allocated to the experimental condition will be asked to complete a Goals Form at the start of every session. This may then form the basis for the evolving clinical dialogue.

Clients allocated to the control condition will begin each session as they would normally do.

At the start of each session, clients in both conditions will be asked to complete the CORE-10.

At the end of therapy, all participants will fill a service satisfaction survey.

Participants in the experimental arm will also take a short quantitative questionnaire to assess the helpfulness of the CORE-10 and the Goals Form.

In addition, a random selection of participants in the experimental arm of the study will be invited back to meet with a researcher to participate in a Qualitative Interview. This will focus on their experience of using the Goals Form, and the ways in which it may, or may not, have been helpful in their therapeutic work.

ELIGIBILITY:
Inclusion Criteria:

* All clients referred for counselling in the service.

Exclusion Criteria:

* Service users who do not understand verbal and written communication in English

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-10-19 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
CORE-10 | 5 minutes

SECONDARY OUTCOMES:
Service satisfaction survey | 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Mick Cooper, D. Phil., Study Director — Professor of Counselling Psychology
Locations (1):
- Tower Hamlets Mind, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anker MG, Duncan BL, Sparks JA. Using client feedback to improve couple therapy outcomes: a randomized clinical trial in a naturalistic setting. J Consult Clin Psychol. 2009 Aug;77(4):693-704. doi: 10.1037/a0016062. PMID 19634962
- [Background] Connell J, Barkham M, Stiles WB, Twigg E, Singleton N, Evans O, Miles JN. Distribution of CORE-OM scores in a general population, clinical cut-off points and comparison with the CIS-R. Br J Psychiatry. 2007 Jan;190:69-74. doi: 10.1192/bjp.bp.105.017657. PMID 17197659
- [Background] Duncan BL, Reese RJ. The Partners for Change Outcome Management System (PCOMS) revisiting the client's frame of reference. Psychotherapy (Chic). 2015 Dec;52(4):391-401. doi: 10.1037/pst0000026. PMID 26641369
- [Result] Farr, J., Di Malta, G. S., & Cooper, M. (2020). Pilot Randomised Controlled Trial of Counselling in a Community Mental Health Setting: Pitfalls and Learnings. Counselling and Psychotherapy Research, 20, 3-8. https://doi.org/10.1002/capr.12262